CLINICAL TRIAL: NCT06449807
Title: Effects of Crossover Point Exercise on Depression, Anxiety and Stress in Chinese Postmenopausal Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ECPEDASCPW
Record Dates: First submitted 2024-02-21; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-02

CONDITIONS: Mental Health
Keywords: Mental health; Sleep quality; Exercise; Body composition; Body image
MeSH Terms: conditions — Psychological Well-Being; Sleep Initiation and Maintenance Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- crossover point intensity exercise (Active Comparator)
  Interventions: Behavioral: crossover point intensity exercise
- No Intervention (No Intervention)

INTERVENTIONS:
Behavioral: crossover point intensity exercise — crossover point intensity exercise
  Arms: crossover point intensity exercise

SUMMARY:
To analyze the effects of the Crossover Point (COP) Exercise Program on Chinese postmenopausal women.

DETAILED DESCRIPTION:
This is a randomized clinical trial of single-blind with 2 arms (control group and experimental group), in which a pre-treatment-posttest design has been used.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women without incapacitating chronic disease or contraindications to exercise
* baseline mental health
* no severe chronic diseases or exercise contraindications
* ability to understand the research details and voluntarily sign the informed consent form.

Exclusion Criteria:

* Women with undetermined menopause；
* BMI <18.5 kg/m2 or BMI >28 kg/m2
* uncontrolled hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >110 mmHg)
* life-threatening illness with a prognosis of <5 years
* currently receiving estrogen therapy
* currently taking medication that may affect psychological testing
* contraindications to exercise

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
DASS-21 (Depression Anxiety Stress Scale-21) | At the beginning-at three months.
  The scale has 21 questions that cover a wide range of symptoms of depression, anxiety, and stress. Each of the questions was stated in the first person, assertive tone, and required the participants to grade on a 4-point scale their experiences with a score of 0 (did not apply to me at all), 1 (applied to me to some degree or some of the time), 2 (applied to me to a considerable degree or a good part of the time), and 3 (applied to me very much or most of the time). The higher value represents a worse result.

SECONDARY OUTCOMES:
Body Mass Index (BMI ) | At the beginning-at three months.
  Is calculated from the formula, Weight (kg) / Height2 (m2), whose unit is kg/m2. It is a rough indicator of total body fat.
Body Image States Scale (BISS) | At the beginning-at three months.
  The BISS contains six items that assess different aspects of body image such as physical appearance, body size and shape, body weight, and attractiveness, as well as concerns about how one looks relative to others. Participants were instructed to complete the questionnaire describing ''How are you feeling right now?'' A higher score represents higher body image satisfaction. The BISS is an internally consistent scale, and construct validity has been confirmed.
Body Appreciation Scale-2 (BAS-2) | At the beginning-at three months.
  The BAS-2 used in this study is the version revised by Swami et al., it comprises a total of 10 items, scored using a Likert five-point scale, corresponding to the options "Never, Rarely, Sometimes, Often, Always," with each item scored from 1 to 5 points. A higher score indicates a stronger appreciation of one's own body.
The Meaning in Life Questionnaire (MLQ) | At the beginning-at three months.
  A reliable, valid and practical screening tool for identifying and quantifying Meaning in Life.
The Subjective Happiness Scale (SMS) | At the beginning-at three months.
  Questionnaire that evaluates the subjective happiness.
Body composition | At the beginning-at three months.
  Body composition indicators analysis was assessed using DXA. Body compositon indicators include: fat mass，lean body mass，percentage of body fat.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Sports Medicine and Rehabilitation, Beijing Sport University, Beijing, China